CLINICAL TRIAL: NCT01718444
Title: Optimizing Fertility Treatment in Women With Polycystic Ovary Syndrome (PCOS) - A Randomized Controlled Trial: The Role of Progestin-induced Endometrial Shedding in PCOS (PIES in PCOS)
Brief Title: Progestin-induced Endometrial Shedding in PCOS (The PIES in PCOS Study)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The primary investigator moved from academic practice to join a private group, and could not get any one to take over as PI for the study.
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Albert Asante, MD MPH, Assistant Professor of Obstetrics-Gynecology, Consultant in Reproductive Endocrinology and Infertility, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-1070
Record Dates: First submitted 2012-10-19; First posted 2012-10-31 (Estimated); Results first posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Polycystic Ovary Syndrome; Infertility
Keywords: PCOS; Polycystic ovary syndrome; Infertility; Anovulation; Clomiphene citrate; Clomid; Progestin; Provera; Progesterone; Endometrial shedding
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility; Anovulation | interventions — Progestins; Medroxyprogesterone Acetate; Clomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (No PIES) (Experimental): Subjects randomized to this group will receive clomiphene citrate (CC) without using progestin throughout their treatment course.
  * CC 50 mg oral for 5 days ("Days 3-7")
  * If no ovulation, CC 100 mg for 5 days ("Days 12-16")
  * If no ovulation, CC 150 mg for 5 days ("Day 21-25")
  * Exit study if no response to 150 mg CC, or if no pregnancy after 5 ovulatory cycles
  Interventions: Drug: Clomiphene Citrate
- Group B (PIES Group) (Active Comparator): Women randomized to this group will receive progestin to induce endometrial shedding before starting any doses of clomiphene citrate (CC)
  * Progestin 10 mg oral for 10 days to induce endometrial shedding (PIES)
  * CC 50 mg oral for 5 days (Day 3-7)
  * If no ovulation, progestin 10 mg for 10 days to induce endometrial shedding (starting on CD28) and CC 100 mg x 5 days, starting on day 3 of induced menses
  * If no ovulation, progestin 10 mg for 10 days to induce endometrial shedding, and CC 150 mg for 5 days
  * Exit study if no response to 150 mg CC, or if no pregnancy after 5 ovulatory cycles
  Interventions: Drug: Progestin; Drug: Clomiphene Citrate

INTERVENTIONS:
Drug: Progestin
  Other Names: Provera; Medroxyprogesterone acetate
  Arms: Group B (PIES Group)
Drug: Clomiphene Citrate
  Other Names: Clomid

SUMMARY:
Progestin-induced endometrial shedding (PIES) followed by clomiphene citrate is fertility treatment of choice in anovulatory women with polycystic ovary syndrome (PCOS). However, some preliminary data suggest that skipping PIES could result in a higher live birth rate. The investigators are performing the first randomized controlled trial to find out if skipping the use of progestin during fertility treatment of anovulatory PCOS women is associated with improved pregnancy and live birth rates compared to the traditional approach of using progestin prior to use of clomiphene citrate.

DETAILED DESCRIPTION:
This is a prospective randomized trial of clomiphene citrate (CC) preceded by progestin-induced endometrial shedding (PIES) vs CC without PIES in the treatment of infertility in patients with PCOS, for up to 5 treatment cycles.

Participants will be randomized to receive either progestin followed by CC starting on day 3 of the induced menses, or CC without induced menses. Study participants will be monitored at regular 2 to 4 wks intervals for response to medication using ultrasound and hormonal parameters. The maximum dose of CC will not exceed 750 mg/cycle. Treatment will not exceed 5 ovulatory cycles. Participants who are resistant to 150 mg of CC will exit the study.

170 anovulatory PCOS women actively seeking pregnancy, aged 18 through 40 years will be enrolled and randomized in a 1:1 treatment ratio into the two study arms. Anovulation will be the only infertility factor in all patients.

ELIGIBILITY:
Inclusion

* Women aged 18 - 40, desiring pregnancy
* Established diagnosis of PCOS confirmed by the Rotterdam criteria
* Oligo or anovulatory, with menstrual cycles > 35 days apart or less than 9 menstrual cycles per year
* Normal vaginal ultrasound with endometrial stripe < 12 mm
* Normal thyroid stimulating hormone (TSH) within past one year
* Normal prolactin (PRL) within past one year
* For women with previous successful Clomid treatment, a washout period of at least 2 months is required

Exclusion

* Regular menstrual cycles occurring less than 35 days apart
* Evidence of other infertility factors such as endometriosis, tubal factor or male infertility
* Prior unsuccessful Clomiphene citrate ovulation cycles
* Abnormal vaginal ultrasound findings such as endometrial polyps, submucous myomas, synechiae
* Uterine anomaly such as unicornuate or bicornuate uterus
* Presence of hydrosalpinx
* Evidence of active endocrinopathy, such as thyroid disorder or hyperprolactinemia
* Partner with abnormal semen analysis (count < 15 million sperm /ml)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2015-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Asante, MD, MPH, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated and data cannot be retrieved as the software where data has been stored has been upgraded. We have exhausted efforts to retrieve the data from this software and no study data are available.
Groups:
- Group A (No PIES): Subjects randomized to this group will receive clomiphene citrate (CC) without using progestin throughout their treatment course.
  * CC 50 mg oral for 5 days ("Days 3-7")
  * If no ovulation, CC 100 mg for 5 days ("Days 12-16")
  * If no ovulation, CC 150 mg for 5 days ("Day 21-25")
  * Exit study if no response to 150 mg CC, or if no pregnancy after 5 ovulatory cycles
  Clomiphene Citrate
- Group B (PIES Group): Women randomized to this group will receive progestin to induce endometrial shedding before starting any doses of clomiphene citrate (CC)
  * Progestin 10 mg oral for 10 days to induce endometrial shedding (PIES)
  * CC 50 mg oral for 5 days (Day 3-7)
  * If no ovulation, progestin 10 mg for 10 days to induce endometrial shedding (starting on CD28) and CC 100 mg x 5 days, starting on day 3 of induced menses
  * If no ovulation, progestin 10 mg for 10 days to induce endometrial shedding, and CC 150 mg for 5 days
  * Exit study if no response to 150 mg CC, or if no pregnancy after 5 ovulatory cycles
  Progestin
  Clomiphene Citrate
Period: Overall Study
Arm/Group | Group A (No PIES) | Group B (PIES Group)
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated and data cannot be retrieved as the software where data has been stored has been upgraded. We have exhausted efforts to retrieve the data from this software and no study data are available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (No PIES) | Group B (PIES Group) | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous [unit: years] — Population: The study was terminated and data cannot be retrieved as the software where data has been stored has been upgraded. We have exhausted efforts to retrieve the data from this software and no study data are available.
Sex: Female, Male — Population: The study was terminated and data cannot be retrieved as the software where data has been stored has been upgraded. We have exhausted efforts to retrieve the data from this software and no study data are available

OUTCOME MEASURES:

1. Primary Outcome: Live Birth
Description: Delivery of a viable infant after 24 weeks of pregnancy
Time Frame: Within 36 weeks of a positive pregnancy test
Population: as for baseline characteristics
Arm/Group | Group A (No PIES) | Group B (PIES Group)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The study was terminated and data cannot be retrieved as the software where data has been stored has been upgraded. We have exhausted efforts to retrieve the data from this software and no study data are available.
Arm/Group | Group A (No PIES) | Group B (PIES Group)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study was terminated and data cannot be retrieved as the software where data has been stored has been upgraded. We have exhausted efforts to retrieve the data from this software and no study data are available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No